CLINICAL TRIAL: NCT01423149
Title: A Phase II, Dose Ranging, Multi-Center Study to Evaluate the Safety and Efficacy of Combretastatin A4 Phosphate for Treating Subfoveal Choroidal Neovascularization in Subjects With Pathologic Myopia
Brief Title: Safety and Efficacy Study of Combretastatin A4 Phosphate to Treat Patients With Choroidal Neovascularization Secondary to Pathologic Myopia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mateon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMD-213
Record Dates: First submitted 2011-08-22; First posted 2011-08-25 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Choroidal Neovascularization; Myopia, Degenerative
Keywords: subfoveal choroidal neovascularization; pathologic myopia
MeSH Terms: conditions — Choroidal Neovascularization; Myopia, Degenerative | interventions — fosbretabulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 36 mg/m2 Combretastin A-4 Phosphate (Experimental)
  Interventions: Drug: Combretastatin A-4 Phosphate
- 45 mg/m2 Combretastatin A-4 Phosphate (Experimental)
  Interventions: Drug: Combretastatin A-4 Phosphate
- 27 mg/m2 Combretastatin A-4 Phosphate (Experimental)
  Interventions: Drug: Combretastatin A-4 Phosphate

INTERVENTIONS:
Drug: Combretastatin A-4 Phosphate — Combretastatin A-4 Phosphate is administered on Day 0 and Day 7 (+/- 2 days). If the treating ophthalmologist notes any leakage from CNV in the study eye on a fluorescein angiography during the study or an increase in subretinal fluid on an optical coherence tomography measurement, retreatment with Combretastatin A-4 Phosphate is recommended with up to 3 additional treatments. The retreatment visit(s) could occur during a scheduled visit or at an additional visit 1 week after a regular study visit. A post-retreatment follow-up visit is necessary.
  Other Names: CA4P; fosbretabulin

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of 3 dose groups (27, 36 and 45 mg/m2) of Combretastatin A-4 Phosphate for the treatment of subfoveal choroidal neovascularization in subjects with pathologic myopia.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Be able and willing to follow instructions
* Age 18 to 50 years old (inclusive)
* Have area of CNV within 50 um or under the geometric center of the foveal avascular zone Have greatest linear dimension of lesion 5,400 um or less, with >/=50.0% of the lesion composed of CNV (features which obscure the boundaries of the CNV such as blood, serous pigment epithelial detachment or blocked fluorescence must occupy <50.0%) as confirmed by Doheny Image Reading Center (DIRC)
* Have best corrected distance visual acuity (ETDRS) of 20/20 to 20/200 (LogMAR +0.0 to 1.0), inclusive in the qualifying eye(s)
* Have pathologic myopia presenting - 6.0 diopters or more correction required OR an axial length of the >/= 26.5 mm
* Be able and willing to avoid any medication that the investigator feels may interfere with the study
* If female and of childbearing potential, agree to submit a sample for pregnancy testing and have a negative pregnancy test within 1 day prior to each treatment. Females are considered of childbearing potential unless they are surgically sterile or post-menopausal for 12 months. Females of childbearing potential must agree to an approved form of contraception for the duration of the study.

Exclusion Criteria:

* Have contraindications, allergies or sensitivity to the use of the study medications
* Have clinical signs or symptoms, in the opinion of the investigator, that may interfere with the study
* Features of any condition other than pathologic myopia associated with CNV, such as age-related macular degeneration
* Have a tear of the retinal pigmented epithelium
* Have undergoing ocular therapy/surgery or major surgery in the last 3 months or have any surgeries planned during the study period
* Have any significant illness or condition, ocular or systemic that could, in the opinion of the investigator, be expected to interfere with the study
* Have angina (stable or severe, even if controlled with medications), 6 months S/P myocardial infarction ,congestive heart failure, history of or presence of any clinically significant supraventricular or ventricular arrhythmias or syncope episodes
* Have ECG with QTc >450 msdec or other clinically significant abnormalities such as left bundle branch block, left ventricular hypertrophy, etc.
* Have uncontrolled QTc prolongation
* Take any drugs known to prolong the QTc interval however subject can remain eligible if a non-QTc substitute can be administered
* Have uncontrolled hypertension (defined as blood pressure consistently greater than 150/100 mm Hg irrespective of medication)
* Uncontrolled hypokalemia and/or hypomagnesemia
* Have symptomatic peripheral vascular disease or cerebrovascular disease
* Have psychiatric disorders or other conditions rendering subjects incapable of complying with the requirements of the protocol
* Be receiving concurrent hormonal therapy with exception of Gonadotropin-releasing hormone agonists in subjects with hormone refractory prostate cancer, hormone replacement therapy, oral contraceptive, and megestrol acetate used for anorexia/cachexia
* Be receiving anticoagulation with warfarin, heparin or low molecular weight heparin other than low dose (1 mg) warfarin for maintenance of Hickman line patency
* Be a woman who is currently pregnant, nursing, or planning a pregnancy; or woman who has a positive pregnancy test
* Have participated in an investigational drug or device trial within 30 days of entering the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2005-03; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity line change from baseline at 3-month following | from baseline to 3 months
Visual acuity response category at 3-month follow-up | from baseline to 3 months

SECONDARY OUTCOMES:
Visual acuity line change from baseline at 1 month follow-up | from baseline to 1 month
Visual acuity response category at 1 month follow-up | from baseline to 1 month
Number of patients with treatment emergent adverse events | from first dose of study drug to 30 days after last dose of study drug

REFERENCES:
- [Derived] Giri P, Batra PJ, Kumari A, Hura N, Adhikary R, Acharya A, Guchhait SK, Panda D. Development of QTMP: A promising anticancer agent through NP-Privileged Motif-Driven structural modulation. Bioorg Med Chem. 2023 Nov 15;95:117489. doi: 10.1016/j.bmc.2023.117489. Epub 2023 Oct 5. PMID 37816266